CLINICAL TRIAL: NCT05246280
Title: Evaluation of Tc 99m Tilmanocept Imaging for the Early Prediction of Anti-TNFα Therapy Response in Patients With Moderate to Severe Active Rheumatoid Arthritis (RA)
Brief Title: Tc 99m Tilmanocept Imaging for Early Prediction of Anti-TNFα Therapy Response in Moderate to Severe Active RA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-33
Record Dates: First submitted 2021-12-16; First posted 2022-02-18 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Tilmanocept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Candidates for initiation of anti-TNFα bDMARD therapy (Experimental): All subjects will be candidates for initiation of, or change to, a new anti-TNFα bDMARD for RA treatment.
  Interventions: Drug: TC99m-tilmanocept

INTERVENTIONS:
Drug: TC99m-tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: tilmanocept; Lymphoseek

SUMMARY:
This study will confirm the ability of Tc 99m tilmanocept imaging to predict clinical response in individuals with RA who are beginning anti-TNFα therapy.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter study designed to evaluate the early predictive capacity of Tc 99m tilmanocept planar imaging for downstream clinical response(s) in individuals with moderate to severe RA who are candidates for change in anti-TNFα therapy. Temporal (Baseline to 5 week) differences in quantitative imaging will be correlated with longitudinal (Baseline to 12- and 24-week) assessments of clinical RA outcomes to evaluate the clinical utility of Tc 99m tilmanocept for the expedited evaluation of antirheumatic treatment efficacy when compared with longitudinal assessments in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
2. The subject is at least 18 years of age and was ≥ 18 years of age at the time of RA diagnosis.
3. The subject is a candidate for initiation of, or change to, a new anti-TNFα bDMARD therapy.
4. The subject has RA as determined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria (score of ≥ 6/10).
5. The subject has moderate to severe RA as determined by a 28-joint disease activity score (DAS28) of ≥ 3.2 (includes the Erythrocyte Sedimentation Rate [ESR] test and Visual Analog Scale [VAS]).
6. Subjects receiving traditional DMARDs must have been on therapy for ≥ 90 days and at a stable dose for ≥ 30 days prior to the first imaging visit (Day 0).
7. Subjects receiving bDMARD or janus kinase (JAK) inhibitor therapy must have been at a stable dose > 60 days prior to the first imaging visit (Day 0).
8. If the subject is receiving NSAIDS (nonsteroidal anti-inflammatory drug) or oral corticosteroids, the dose has been stable for > 28 days prior to the first imaging visit (Day 0). The corticosteroid dose must be ≤ 10 mg/day of prednisone or an equivalent steroid dose.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject size or weight is not compatible with imaging per the investigator.
3. The subject is currently receiving radiation therapy or chemotherapy or has received radiation or chemotherapy within the past 5 years.
4. The subject has an active malignancy or a history of malignancy within the past 5 years.
5. The subject has had a finger, hand, and/or wrist amputation or hand or wrist joint arthroplasty.
6. The subject has renal insufficiency as demonstrated by a glomerular filtration rate of < 60 mL/min.
7. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than 2 times the upper limit of normal.
8. The subject has any severe, acute, or chronic medical conditions and/or psychiatric conditions and/or laboratory abnormalities that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration that would deem the subject inappropriate for study participation.
9. The subject has a history of hypersensitivity reactions to TNF-inhibitors.
10. The subject has a known allergy to or has had an adverse reaction to dextran exposure.
11. The subject has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration at the first imaging visit (Day 0).
12. The subject has received intra-articular corticosteroid injections ≤ 8 weeks prior to the first imaging visit (Day 0).
13. The subject has received any radiopharmaceutical within 7 days or 10 half-lives prior to the administration of Tc 99m tilmanocept at the first imaging visit (Day 0).
14. The subject has heart failure [New York Heart Association (NYHA) Class III-IV], a demyelinating disorder, or a chronic/latent infection [e.g., +Purified Protein Derivative (PPD) test, Human Immunodeficiency Virus (HIV), Hepatitis B].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (13):
- United States (13):
  - Attune Health Research, Beverly Hills, California
  - University of California, San Francisco, San Francisco, California
  - Highlands Advanced Rheumatology and Arthritis Center, Avon Park, Florida
  - Believe Clinical Trials, Coral Springs, Florida
  - Nouvelle Clinical Research, Cutler Bay, Florida
  - Vida Clinical Research, Kissimmee, Florida
  - Life Clinical Trials, Margate, Florida
  - D&H National Research Centers, Inc, Miami, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Physician Research Collaboration, Lincoln, Nebraska
  - Essential Medical Research, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis and Osteoporosis Center of Coastal Bend, Corpus Christi, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Started | 169
Completed | 169
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 128
  >=65 years | 41
Age, Continuous [Mean (Full Range); unit: years] | 59.2 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 146
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 169

OUTCOME MEASURES:

1. Primary Outcome: Specificity of Tilmanocept Uptake Value (TUV)
Description: Specificity of the change in TUVglobal with bucketing from baseline to 5 weeks after a change in anti-TNFα therapy (ΔTUVglobal[5w] with bucketing) with respect to ACR50 at week 24 after the change in therapy.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Sensitivity of Tilmanocept Uptake Value (TUV)
Description: Sensitivity of the change in TUVglobal with bucketing from baseline to 5 weeks after change in anti-TNFα therapy (ΔTUVglobal[5w] with bucketing) with respect to ACR50 at week 24 after the change in therapy.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Negative Predictive Value (NPV) of TUV Baseline at Week 24
Description: NPV of TUV global obtained at baseline (TUVglobal[b]) with respect to ACR50 at week 24 after change in anti-TNFα therapy
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Sensitivity and Specificity of ΔTUVglobal[5w] With Bucketing With Respect to ACR50 at Week 12
Description: Concordance of ΔTUVglobal[5w] with bucketing and ACR50 at week 12, evaluated using sensitivity and specificity.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: NPV, and PPV, and OA of ΔTUVglobal[5w] With Bucketing With Respect to ACR50 at Weeks 12 and 24
Description: Concordance of ΔTUVglobal[5w] (with bucketing) and clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI©. Concordance between ΔTUVglobal[5w] and the clinical criteria will be evaluated using NPV, PPV and overall accuracy.
Time Frame: up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Negative Predictive Value (NPV) of TUV Baseline at Week 12
Description: Negative predictive value (NPV) of TUVglobal obtained at baseline (TUVglobal[b]) with respect to ACR50 at week 12
Time Frame: up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Concordance of TUV Baseline and Change in Clinical Disease Activity Index (CDAI), 28-joint Count Disease Activity Score (DAS28), and American College of Rheumatology (ACR) Response Criteria
Description: TUVglobal[b] and response to new anti-TNFα bDMARD therapy defined by the change from baseline (CFB) of CDAI to 12 +/- 1 weeks and 24 +/- 1 weeks, by the CFB of DAS28 to 12 +/- 1 weeks and 24 +/- 1 weeks and by the CFB in each of the ACR Response Criteria components at 12 +/- 1 weeks and at 24 +/- 1 weeks.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

8. Secondary Outcome: Concordance of TUV Baseline to Week 5 and Change in Clinical Disease Activity Index (CDAI)
Description: ΔTUVglobal[5w] and response to new anti-TNFα bDMARD therapy defined by the CFB of CDAI to 12 +/- 1 weeks and 24 +/- 1 weeks.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

9. Secondary Outcome: Concordance of TUV Baseline to Week 5 and Clinical Disease Activity Index (CDAI),28-joint Count Disease Activity Score (DAS28), and American College of Rheumatology (ACR) Response Criteria
Description: Concordance of ΔTUVglobal[5w] (without bucketing) and clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI©. Concordance between ΔTUVglobal[5w] and the clinical criteria will be evaluated using NPV, PPV, sensitivity, specificity, and overall accuracy.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

10. Secondary Outcome: Concordance of TUV Baseline to Week 12 and Clinical Disease Activity Index (CDAI),28-joint Count Disease Activity Score (DAS28), and American College of Rheumatology (ACR) Response Criteria
Description: Concordance of ΔTUVglobal[12w] and change in clinical criteria, including ACR Response Criteria, CDAI, DAS28, and HAQ-DI©. Concordance between ΔTUVglobal[12w] and the clinical criteria will be evaluated using NPV, PPV, sensitivity, specificity, and overall accuracy.
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

11. Secondary Outcome: Correlation of TUV Baseline to Week 5 and ACR Response Criteria Components
Description: Correlation of ΔTUVglobal[5w] and response to new anti-TNFα bDMARD therapy from baseline to 24 +/- 1 weeks defined by the changes from baseline in each of the ACR Response Criteria components, including:
  * Tender joint count (TJC)
  * Swollen joint count (SJC)
  * Patient assessment of global disease activity
  * Rheumatologist assessment of global disease activity
  * Patient assessment of pain
  * Patient assessment of physical function
  * Acute-phase reactant value
Time Frame: Up to 213 days
Population: Data not collected.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 0

12. Secondary Outcome: Safety of IV-administered Tilmanocept Radiolabled With Tc 99m Assessed by AEs
Description: Incidence of AEs related to Tc 99m tilmanocept.
Time Frame: Up to 213 days
Population: All subjects injected with Tc 99m tilmanocept were evaluated.
Measure: Number; unit: Adverse Events
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 169
Adverse Events
  Adverse Events Severity - Mild | 47
  Adverse Events Severity - Moderate | 84
  Adverse Events Severity - Severe | 1
  Adverse Events Relatedness - Possibly Related | 1
  Adverse Events Relatedness - Probably Not Related | 1
  Adverse Events Relatedness - Definitely Not Related | 130

13. Secondary Outcome: Safety of IV-administered Tilmanocept Radiolabled With Tc 99m Assessed by Number of Participants With Changes Over Time in Clinical Laboratory Tests
Description: Number of participants with changes over time in clinical laboratory tests (hematology, serum chemistry, urinalysis, and RA panel).
Time Frame: Up to 213 days
Population: All subjects injected with Tc 99m tilmanocept were evaluated.
Measure: Number; unit: Participants
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 169
Participants | 2

14. Secondary Outcome: Safety of IV-administered Tilmanocept Radiolabled With Tc 99m Assessed by Number of Participants With Changes Over Time in ECG Parameters
Description: Number of participants with changes over time in ECG parameters (PRS Interval, QRS Duration, QT Interval, and QTc Interval).
Time Frame: Up to 213 days
Population: All subjects injected with Tc 99m tilmanocept were evaluated.
Measure: Number; unit: participants
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 169
participants | 2

15. Secondary Outcome: Safety of IV-administered Tilmanocept Radiolabled With Tc 99m Assessed by Number of Participants With Changes Over Time in Vital Signs
Description: Number of participants with changes over time in vital signs (blood pressure, heart rate, respiratory rate, and temperature).
Time Frame: Up to 213 days
Population: All subjects injected with Tc 99m tilmanocept were evaluated.
Measure: Number; unit: participants
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
Number analyzed (Participants) | 169
participants | 9

ADVERSE EVENTS:
Time Frame: Up to 213 days.
Arm/Group | Candidates for Initiation of Anti-TNFα bDMARD Therapy
All-Cause Mortality (participants affected / at risk) | 0/169
Serious Adverse Events (participants affected / at risk) | 5/169
Other Adverse Events (participants affected / at risk) | 0/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candidates for Initiation of Anti-TNFα bDMARD Therapy (N=169)
scalp laceration (Skin and subcutaneous tissue disorders) | 1 (1) — The sbj, a 78-year-old female, fell from a ladder and was hospitalized due to a scalp laceration. The scalp laceration was serious due to hospitalization, moderate in intensity, and unexpected. All events were reported as definitely not related.
Blunt abdominal trauma (Social circumstances) | 1 (1) — The subject, a 63-year-old female, was in a motor vehicle accident and hospitalized due to blunt abdominal trauma, abdominal ecchymosis and right index finger pain. All events were reported as definitely not related.
snycope (Cardiac disorders) | 1 (1) — The subject, a 70-year-old female, was hospitalized due to syncope. It was reported as definitely not related to the investigational drug or procedure.
acute appendicitis (General disorders) | 1 (1) — The subject, a 74-year-old female, was hospitalized due to appendicitis perforated on 04 July 2023. It was reported as definitely not related to the investigational drug or procedure.
Non-Cardiac Atypical Chest Pain (Cardiac disorders) | 1 (1) — The subject, a 57-year-old female, was hospitalized due to noncardiac atypical chest pain on 02 March 2023. It was reported as definitely not related to the investigational drug or procedure.

LIMITATIONS AND CAVEATS:
Available data from this trial was being presented as an abbreviated clinical study report to the FDA under the IND as not all efficacy analyses were completed. The trail was halted before completion; therefore tables, listings, and figures were not generated. All available safety data has been presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement states that no publications will be made unless approval by the sponsor is granted.

DOCUMENTS (3):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05246280/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT05246280/SAP_002.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT05246280/ICF_001.pdf